CLINICAL TRIAL: NCT05049499
Title: Long-term Academic and Psychosocial Impact of Child's Sleep: Parental Influences
Status: Active, not recruiting | Type: Observational
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, June Chi Yan Lo, Assistant Professor, National University of Singapore
Other Study IDs: LAPICS
Record Dates: First submitted 2021-08-30; First posted 2021-09-20 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Parents; School-age Children; Sleep; Academic Achievements; Mental Well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The proposed longitudinal project aims to understand parental influences on children's sleep and will investigate the effect of sleep-related parental factors - (1) parents' value of their children's sleep relative to other activities, (2) parental involvement in setting children's sleep habits and enforcing good sleep hygiene, and (3) parent's own sleep habits - on school-age children's sleep, mental health, socio-emotional resilience, and academic/cognitive performance. It will also investigate the impact of social economic status on these sleep -related parental factors.

DETAILED DESCRIPTION:
Parents can influence their children's sleep in various ways. However, existing studies on parental factors of school-aged children's sleep have seldom moved beyond sleep hygiene and the relationships between parent and child's sleep patterns. A potential factor that has been overlooked is parents' value of their children's sleep - whether they value their children's sleep and prioritise it over other activities, e.g. studying or watching TV. Another variable to consider is the social economic status (SES) of the household, which can influence these parental factors.

The proposed longitudinal project will investigate the impact of SES on several sleep-related parental factors and the effects these parental factors have on children's sleep, mental health, socio-emotional resilience, and academic/cognitive performance. The project will involve school-age children in Singapore (baseline age: 7-12 years) at two time points, time 1 (T1) and time 2 (T2), one year apart.

At each timepoint, children's sleep will be assessed with actigraphy for 1 school week. This will be followed by a lab visit during which sleep-related parental factors, as well as the children's sleep, academic and cognitive performance, socio-emotional resilience, and mental health will be assessed. Lab visits will be scheduled at the end of the school week in the morning and early afternoon so that neurobehavioural functions can be captured during typical school hours.

Investigators hypothesise that parents from low SES households will value their child's sleep less, and therefore, allow their child to trade a larger amount of sleep for other activities. Parents from low SES households will also enforce good sleep hygiene less, and sleep less themselves. Children from low SES households will thus have shorter sleep duration, more sleep disturbance, poorer mental health, poorer socio-emotional resilience, and poorer academic and cognitive performance.

ELIGIBILITY:
Inclusion Criteria:

* Is aged between 7 and 12 years
* Is a Singaporean
* Is English-speaking
* Is not on any long-term medications
* Has no known medical conditions that could affect sleep (e.g. asthma)
* Has no history of psychiatric or neurological disorders
* Has no history of sleep problems / disorders

Exclusion Criteria:

The reverse of the inclusion criteria

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: School-age children (between 7 and 12 years old) in Singapore
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of minutes of sleep allowed to be traded for studying on weekdays | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for studying (including homework and tuition) on weekdays
Number of minutes of sleep allowed to be traded for studying on weekdays | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for studying (including homework and tuition) on weekdays
Number of minutes of sleep allowed to be traded for studying on weekends | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for studying (including homework and tuition) on weekends
Number of minutes of sleep allowed to be traded for studying on weekends | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for studying (including homework and tuition) on weekends
Number of minutes of sleep allowed to be traded for co-/extra-curricular activities on weekdays | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for co-/extra-curricular activities on weekdays
Number of minutes of sleep allowed to be traded for co-/extra-curricular activities on weekdays | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for co-/extra-curricular activities on weekdays
Number of minutes of sleep allowed to be traded for co-/extra-curricular activities on weekends | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for co-/extra-curricular activities on weekends
Number of minutes of sleep allowed to be traded for co-/extra-curricular activities on weekends | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for co-/extra-curricular activities on weekends
Number of minutes of sleep allowed to be traded for interacting face to face with family / friends on weekdays | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for interacting face to face with family / friends on weekdays
Number of minutes of sleep allowed to be traded for interacting face to face with family / friends on weekdays | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for interacting face to face with family / friends on weekdays
Number of minutes of sleep allowed to be traded for interacting face to face with family / friends on weekends | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for interacting face to face with family / friends on weekends
Number of minutes of sleep allowed to be traded for interacting face to face with family / friends on weekends | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for interacting face to face with family / friends on weekends
Number of minutes of sleep allowed to be traded for social media on weekdays | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for social media on weekdays
Number of minutes of sleep allowed to be traded for social media on weekdays | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for social media on weekdays
Number of minutes of sleep allowed to be traded for social media on weekends | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for social media on weekends
Number of minutes of sleep allowed to be traded for social media on weekends | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for social media on weekends
Number of minutes of sleep allowed to be traded for gaming on weekdays | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for gaming on weekdays
Number of minutes of sleep allowed to be traded for gaming on weekdays | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for gaming on weekdays
Number of minutes of sleep allowed to be traded for gaming on weekends | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for gaming on weekends
Number of minutes of sleep allowed to be traded for gaming on weekends | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for gaming on weekends
Number of minutes of sleep allowed to be traded for watching TV / videos on weekdays | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for watching TV / videos on weekdays
Number of minutes of sleep allowed to be traded for watching TV / videos on weekdays | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for watching TV / videos on weekdays
Number of minutes of sleep allowed to be traded for watching TV / videos on weekends | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for watching TV / videos on weekends
Number of minutes of sleep allowed to be traded for watching TV / videos on weekends | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for watching TV / videos on weekends
Number of minutes of sleep allowed to be traded for other activities (non-listed) on weekdays | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for other activities (not already listed above) on weekdays
Number of minutes of sleep allowed to be traded for other activities (non-listed) on weekdays | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for other activities (not already listed above) on weekdays
Number of minutes of sleep allowed to be traded for other activities (non-listed) on weekends | At year 1
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for other activities (not already listed above) on weekends
Number of minutes of sleep allowed to be traded for other activities (non-listed) on weekends | At year 2
  Parents will indicate the number of minutes they allow their child to sleep less in exchange for more time for other activities (not already listed above) on weekends
Parent-set bedtime on weekdays | At year 1
  Parents will indicate whether they allow their children to decide their own bedtimes on weekdays
Parent-set bedtime on weekdays | At year 2
  Parents will indicate whether they allow their children to decide their own bedtimes on weekdays
Parent-set bedtime on weekends | At year 1
  Parents will indicate whether they allow their children to decide their own bedtimes on weekends
Parent-set bedtime on weekends | At year 2
  Parents will indicate whether they allow their children to decide their own bedtimes on weekends
Parent-set wake time on weekdays | At year 1
  Parents will indicate whether they allow their children to decide their own wake times on weekdays
Parent-set wake time on weekdays | At year 2
  Parents will indicate whether they allow their children to decide their own wake times on weekdays
Parent-set wake time on weekends | At year 1
  Parents will indicate whether they allow their children to decide their own wake times on weekends
Parent-set wake time on weekends | At year 2
  Parents will indicate whether they allow their children to decide their own wake times on weekends
Child's usage of electronic device 1 hour before bedtime | At year 1
  Parents will indicate whether their child uses any electronic device 1 hour before going to bed
Child's usage of electronic device 1 hour before bedtime | At year 2
  Parents will indicate whether their child uses any electronic device 1 hour before going to bed
Noise during child's sleep time | At year 1
  Questions include:
  Is your home noisy during his/her sleep time? (Not noisy, A little noisy, Noisy) Does your child take his/her phone into the bedroom close to bed time? (Yes, No, N.A) Does your child put his/her phone on silent mode or switch it off before going to bed? (Yes, No, N.A.)
Noise during child's sleep time | At year 2
  Questions include:
  Is your home noisy during his/her sleep time? (Not noisy, A little noisy, Noisy) Does your child take his/her phone into the bedroom close to bed time? (Yes, No, N.A) Does your child put his/her phone on silent mode or switch it off before going to bed? (Yes, No, N.A.)
Temperature in the bedroom during child's sleep time | At year 1
  Questions include:
  Is any of the following cooling devices used in his/her room during his/her sleep time? (Air conditioner, Electric fan, Both air conditioner and electric fan, Neither air conditioner nor electric fan) What is the average temperature of his/her room during his/her sleep time? (°C)
Temperature in the bedroom during child's sleep time | At year 2
  Questions include:
  Is any of the following cooling devices used in his/her room during his/her sleep time? (Air conditioner, Electric fan, Both air conditioner and electric fan, Neither air conditioner nor electric fan) What is the average temperature of his/her room during his/her sleep time? (°C)
Darkness of the bedroom during child's sleep time | At year 1
  Questions include:
  How dark is his/her room during his/her sleep time? (1. Very bright, 2. Moderately bright, 3. Average, 4. Moderately dark, 5. Entirely or almost entirely dark) If your child's bedroom is not completely dark during bedtime, what are the types of light source that are present in his/her bedroom? (The bedroom is completely dark, Room light / Nightlight, Light from another room inside the house, Light from outside the house)
Darkness of the bedroom during child's sleep time | At year 2
  Questions include:
  How dark is his/her room during his/her sleep time? (1. Very bright, 2. Moderately bright, 3. Average, 4. Moderately dark, 5. Entirely or almost entirely dark) If your child's bedroom is not completely dark during bedtime, what are the types of light source that are present in his/her bedroom? (The bedroom is completely dark, Room light / Nightlight, Light from another room inside the house, Light from outside the house)
Child's daily caffeine consumption | At year 1
  Parents will indicate the average amount of caffeine their child typically consumes each day.
Child's daily caffeine consumption | At year 2
  Parents will indicate the average amount of caffeine their child typically consumes each day.
Parents' work schedule assessed by what time parent's leave for work | At year 1
  Parents will report the time they usually leave the house for work.
Parents' work schedule assessed by what time parent's leave for work | At year 2
  Parents will report the time they usually leave the house for work.
Parents' work schedule assessed by what time parent's reach home | At year 1
  Parents will report the time they usually reach home after work.
Parents' work schedule assessed by what time parent's reach home | At year 2
  Parents will report the time they usually reach home after work.
Parents' bedtime on weekdays | At year 1
  Parents will report the time they usually go to bed on weekdays.
Parents' bedtime on weekdays | At year 2
  Parents will report the time they usually go to bed on weekdays.
Parents' bedtime on weekends | At year 1
  Parents will report the time they usually go to bed on weekends.
Parents' bedtime on weekends | At year 2
  Parents will report the time they usually go to bed on weekends.
Parents' wake time on weekdays | At year 1
  Parents will report the time they usually wake up on weekdays.
Parents' wake time on weekdays | At year 2
  Parents will report the time they usually wake up on weekdays.
Parents' wake time on weekends | At year 1
  Parents will report the time they usually wake up on weekends.
Parents' wake time on weekends | At year 2
  Parents will report the time they usually wake up on weekends.
Parents' sleep duration on weekdays | At year 1
  Parents will report their usual sleep duration on weekdays.
Parents' sleep duration on weekdays | At year 2
  Parents will report their usual sleep duration on weekdays.
Parents' sleep duration on weekends | At year 1
  Parents will report their usual sleep duration on weekends.
Parents' sleep duration on weekends | At year 2
  Parents will report their usual sleep duration on weekends.
Child's time in bed as measured by actigraphy | At year 1
  Participants will wear an actiwatch (Actiwatch 2, Philips Respironics) around the wrist of their non-dominant hand for one week during school term. Data will be collected at 30-second resolution.
Child's time in bed as measured by actigraphy | At year 2
  Participants will wear an actiwatch (Actiwatch 2, Philips Respironics) around the wrist of their non-dominant hand for one week during school term. Data will be collected at 30-second resolution.
Child's total sleep time as measured by actigraphy | At year 1
  Participants will wear an actiwatch (Actiwatch 2, Philips Respironics) around the wrist of their non-dominant hand for one week during school term. Data will be collected at 30-second resolution.
Child's total sleep time as measured by actigraphy | At year 2
  Participants will wear an actiwatch (Actiwatch 2, Philips Respironics) around the wrist of their non-dominant hand for one week during school term. Data will be collected at 30-second resolution.
Child's sleep efficiency as measured by actigraphy | At year 1
  Participants will wear an actiwatch (Actiwatch 2, Philips Respironics) around the wrist of their non-dominant hand for one week during school term. Data will be collected at 30-second resolution.
Child's sleep efficiency as measured by actigraphy | At year 2
  Participants will wear an actiwatch (Actiwatch 2, Philips Respironics) around the wrist of their non-dominant hand for one week during school term. Data will be collected at 30-second resolution.
Child's subjective sleep quality | At year 1
  Participants will report their subjective sleep quality using an item modified from the Pittsburgh Sleep Quality Index - "How would you rate the quality of your sleep last night?" ("Very good" / "Fairly good" / "Fairly bad" / "Very bad").
Child's subjective sleep quality | At year 2
  Participants will report their subjective sleep quality using an item modified from the Pittsburgh Sleep Quality Index - "How would you rate the quality of your sleep last night?" ("Very good" / "Fairly good" / "Fairly bad" / "Very bad").
Child's bedtime on weekdays as reported by parents | At year 1
  Parents will report their child's usual bedtime on weekdays.
Child's bedtime on weekdays as reported by parents | At year 2
  Parents will report their child's usual bedtime on weekdays.
Child's bedtime on weekends as reported by parents | At year 1
  Parents will report their child's usual bedtime on weekends.
Child's bedtime on weekends as reported by parents | At year 2
  Parents will report their child's usual bedtime on weekends.
Child's wake time on weekdays as reported by parents | At year 1
  Parents will report their child's usual wake time on weekdays.
Child's wake time on weekdays as reported by parents | At year 2
  Parents will report their child's usual wake time on weekdays.
Child's wake time on weekends as reported by parents | At year 1
  Parents will report their child's usual wake time on weekends.
Child's wake time on weekends as reported by parents | At year 2
  Parents will report their child's usual wake time on weekends.
Child's sleep duration on weekdays as reported by parents | At year 1
  Parents will report their child's usual sleep duration on weekdays.
Child's sleep duration on weekdays as reported by parents | At year 2
  Parents will report their child's usual sleep duration on weekdays.
Child's sleep duration on weekends as reported by parents | At year 1
  Parents will report their child's usual sleep duration on weekends.
Child's sleep duration on weekends as reported by parents | At year 2
  Parents will report their child's usual sleep duration on weekends.
Frequency of child's sleep-related problems | At year 1
  The sum of the reported frequency (0 = never; 1 = < 1 time per month, 2 = 1-2 times per month, 3 = 1-2 times per week, 4 = ≥ 3 times per week) at which their child experiences various sleep-related problems. Statements/questions include:
  Difficulty falling asleep; Anxious or afraid when falling asleep; Repetitive rocking movements or head banging while falling asleep; Startled or jerky movements of body parts while asleep; Sweating frequently during the night; Sudden awakening during sleep; Breathing difficulty during sleep; Mouth breathing during sleep; Breath holding or pausing during sleep; Lips turning blue while asleep; Frequent position changes while asleep Sleeping in prone position with buttocks up and neck extended; Teeth grinding during sleep; Bed wetting during sleep; Sleep talking; Nightmares; Waking up in the early morning and unable to fall back asleep; Dry mouth in the morning; Did he/she have any other sleep problems?
Frequency of child's sleep-related problems | At year 2
  The sum of the reported frequency (0 = never; 1 = < 1 time per month, 2 = 1-2 times per month, 3 = 1-2 times per week, 4 = ≥ 3 times per week) at which their child experiences various sleep-related problems. Statements/questions include:
  Difficulty falling asleep; Anxious or afraid when falling asleep; Repetitive rocking movements or head banging while falling asleep; Startled or jerky movements of body parts while asleep; Sweating frequently during the night; Sudden awakening during sleep; Breathing difficulty during sleep; Mouth breathing during sleep; Breath holding or pausing during sleep; Lips turning blue while asleep; Frequent position changes while asleep Sleeping in prone position with buttocks up and neck extended; Teeth grinding during sleep; Bed wetting during sleep; Sleep talking; Nightmares; Waking up in the early morning and unable to fall back asleep; Dry mouth in the morning; Did he/she have any other sleep problems?
Sustained attention assessed with the 5-minute Psychomotor Vigilance Task | At year 1
  Number of attention lapses (>500ms)
Sustained attention assessed with the 5-minute Psychomotor Vigilance Task | At year 2
  Number of attention lapses (>500ms)
Median reaction time assessed with the 5-minute Psychomotor Vigilance Task | At year 1
  Median reaction time
Median reaction time assessed with the 5-minute Psychomotor Vigilance Task | At year 2
  Median reaction time
Standard deviation of reaction time assessed with the 5-minute Psychomotor Vigilance Task | At year 1
  Standard deviation of reaction time
Standard deviation of reaction time assessed with the 5-minute Psychomotor Vigilance Task | At year 2
  Standard deviation of reaction time
Child's academic performance | At year 1
  Parents will respond to two questions: "how well do you feel your child is performing at school" and "combining across all subjects, what is your child's typical overall grade in school".
Child's academic performance | At year 2
  Parents will respond to two questions: "how well do you feel your child is performing at school" and "combining across all subjects, what is your child's typical overall grade in school".
Child's daytime sleepiness | At year 1
  Child's daytime sleepiness will be indicated by the total score of the Pediatric Daytime Sleepiness Scale.
Child's daytime sleepiness | At year 2
  Child's daytime sleepiness will be indicated by the total score of the Pediatric Daytime Sleepiness Scale.
Child's socio-emotional resilience assessed by the child's ability to accept responsibility and to regulate his/her emotion | At year 1
  Parents will fill in the Social-Emotional Assets and Resilience Scales-Parent form (SEARS-P), which consists of 39 items. The total score of each subscale will be used to respectively indicate the child's ability to regulate his / her emotion and accept responsibility, make friends, and empathise.
Child's socio-emotional resilience assessed by the child's ability to accept responsibility and to regulate his/her emotion | At year 2
  Parents will fill in the Social-Emotional Assets and Resilience Scales-Parent form (SEARS-P), which consists of 39 items. The total score of each subscale will be used to respectively indicate the child's ability to regulate his / her emotion and accept responsibility, make friends, and empathise.
Child's socio-emotional resilience assessed by the child's ability to make friends | At year 1
  Parents will fill in the Social-Emotional Assets and Resilience Scales-Parent form (SEARS-P), which consists of 39 items. The total score of each subscale will be used to respectively indicate the child's ability to regulate his / her emotion and accept responsibility, make friends, and empathise.
Child's socio-emotional resilience assessed by the child's ability to make friends | At year 2
  Parents will fill in the Social-Emotional Assets and Resilience Scales-Parent form (SEARS-P), which consists of 39 items. The total score of each subscale will be used to respectively indicate the child's ability to regulate his / her emotion and accept responsibility, make friends, and empathise.
Child's socio-emotional resilience assessed by the child's ability to empathise | At year 1
  Parents will fill in the Social-Emotional Assets and Resilience Scales-Parent form (SEARS-P), which consists of 39 items. The total score of each subscale will be used to respectively indicate the child's ability to regulate his / her emotion and accept responsibility, make friends, and empathise.
Child's socio-emotional resilience assessed by the child's ability to empathise | At year 2
  Parents will fill in the Social-Emotional Assets and Resilience Scales-Parent form (SEARS-P), which consists of 39 items. The total score of each subscale will be used to respectively indicate the child's ability to regulate his / her emotion and accept responsibility, make friends, and empathise.
Child's depression symptoms | At year 1
  Parents will report the frequency at which their child experiences each of the 10 depression symptoms on the 25-item Revised Child Anxiety and Depression Scale.
Child's depression symptoms | At year 2
  Parents will report the frequency at which their child experiences each of the 10 depression symptoms on the 25-item Revised Child Anxiety and Depression Scale.
Child's anxiety symptoms | At year 1
  Parents will report the frequency at which their child experiences each of the 15 anxiety symptoms on the 25-item Revised Child Anxiety and Depression Scale.
Child's anxiety symptoms | At year 2
  Parents will report the frequency at which their child experiences each of the 15 anxiety symptoms on the 25-item Revised Child Anxiety and Depression Scale.
Child's internalising behaviour | At year 1
  Parents will complete the Child Behaviour Checklist that assesses their child's internalising behaviour at Time 1
Child's internalising behaviour | At year 2
  Parents will complete the Child Behaviour Checklist that assesses their child's internalising behaviour at Time 2
Child's externalising behaviour | At year 1
  Parents will complete the Child Behaviour Checklist that assesses their child's externalising behaviour at Time 1.
Child's externalising behaviour | At year 2
  Parents will complete the Child Behaviour Checklist that assesses their child's externalising behaviour at Time 2
Child's age | At year 1
  Parents will report child's age at Time 1
Child's age | At year 2
  Parents will report child's age at Time 2
Child's gender | At year 1
  Parents will report child's gender.
Child's ethnicity | At year 1
  Parents will report child's ethnicity.
Parents' age | At year 1
  Parents will report their ages at Time 1
Parents' age | At year 2
  Parents will report their ages at Time 2
Parents' education level | At year 1
  Parents will report their education level at Time 1
Parents' education level | At year 2
  Parents will report their education level at Time 2
Parents' marital status | At year 1
  Parents will report their marital status at Time 1
Parents' marital status | At year 2
  Parents will report their marital status at Time 2
Socioeconomic status assessed by the type of accommodation | At year 1
  Parents will report the type of accommodation they are living in at Time 1
Socioeconomic status assessed by the type of accommodation | At year 2
  Parents will report the type of accommodation they are living in at Time 2
Socioeconomic status assessed by monthly household income | At year 1
  Parents will report their monthly household income at Time 1
Socioeconomic status assessed by monthly household income | At year 2
  Parents will report their monthly household income at Time 2

CONTACTS AND LOCATIONS:
Overall Officials: June Chi Yan Lo, Ph.D., Principal Investigator — National University of Singapore
Locations (1):
- National University of Singapore, Singapore, Singapore